CLINICAL TRIAL: NCT04048564
Title: Observational Study on CML Patients in Any Phase of the Disease Treated With Ponatinib (Iclusig®): A Multicentre, Ambispective Cohort Study
Brief Title: Observational Study on CML Patients in Any Phase of the Disease Treated With Ponatinib (Iclusig®)
Status: Completed | Type: Observational
Sponsor: Incyte BioSciences France (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Other Study IDs: 2017-A01355-48
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Iclusig; ponatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentre ambispective cohort study involving French patients who have started or are receiving for less than 6 months a treatment with ponatinib. This study aims at better qualifying the ponatinib benefit-risk balance in real life and in relation with CML patients' therapeutic history.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a CML in any phase.
* Having initiated for less than six months a treatment with ponatinib.
* The ability to understand the requirements of the study and to comply with the study data collection procedures.

Exclusion Criteria:

* Patients previously treated with investigational ponatinib (within a clinical trial).
* Patients receiving an investigational agent.
* Patients who are pregnant and/or breastfeeding.
* Patients with contraindications for Ponatinib according to Summary of Products Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 public and private French investigative centers of hematology will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
For participants in chronic myeloid leukemia in chronic (CP-CML) phase: Proportion of participants who achieve a major molecular response after the initiation of study treatment | from 24-60 months
  Chronic myeloid leukemia (CML) response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia (Hochhaus et al Leukemia 2020).
For participants in chronic myeloid leukemia in accelerated phase (AP-CML) or chronic myeloid leukemia in blast phase (BP-CML): Proportion of participants who achieve a complete hematologic response | from 24-60 months
  CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.

SECONDARY OUTCOMES:
Proportion of participants in CP-CML phase who achieved complete hematologic response | from 24-60 months
  CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.
Proportion of participants in AP and BP phases who achieved major (complete + partial) cytogenetic response | from 24-60 months
  CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.
Proportion of participants who achieved major molecular response and/or depth molecular response: (MR4 or MR4.5 or MR5) | from 24-60 months
  CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.
Duration of response | from 24-60 months
  Duration of CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.
Time to progression to AP-CML or BP-CML (for those participants not in AP-CML or BP-CML) | from 24-60 months
  Time to progression to AP-CML defined as follows: Blasts in blood or marrow 15%-29%, or blasts plus promyelocytes in blood or marrow > 30%, with blasts < 30%; basophils in blood ≥ 20%; persistent thrombocytopenia (< 100 × 10^9/L) unrelated to therapy; clonal chromosome abnormalities in Ph1 cells (CCA/Ph1), major route, on treatment. Time to progression to BP-CML defined as follows: Blasts in blood or marrow ≥ 30%; extramedullary blast proliferation, apart from spleen.
Dose reduction (after response) in each cohort | from 24-60 months
  Includes level of response at the time of dose reduction and maintenance of response after dose reduction.
Time to response | from 24-60 months
  Time to CML response criteria as defined by the European LeukemiaNet Recommendations for Management of Chronic Myeloid Leukemia.
Rate of progression to accelerated phase (AP-) or blast phase (BP-) CML | from 24-60 months
  Rate of progression to AP- or BP-CML as defined in European LeukemiaNet (ELN) criteria.
Progression-free survival (PFS) | from 24-60 months
  Survival without any progression to AP or BP according to ELN criteria.
Overall survival (OS) | from 24-60 months
  Overall survival defined according to ELN criteria.
Rate of adverse events | from 24-60 months
  Adverse event is any untoward medical occurrence in a patient or clinical study subject administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment.
Rate of discontinuation due to adverse events in each dose cohort | from 24-60 months
  Adverse event is any untoward medical occurrence in a patient or clinical study subject administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment.
Dose reductions (prior to response) in each dose cohort | from 24-60 months
  Reduction in the dose of Iclusig.
Dose interruptions in each dose cohort | from 24-60 months
  Interruption of Iclusig treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ali G. Turnan, MD, PhD, Principal Investigator — Paris Sud University Hospitals-Bicetre
Locations (40):
- France (40):
  - CHU SUD Reunion GHSR, Saint-Pierre, Reunion
  - CHU Amiens-Picardie- Site SUD, Amiens
  - CHU D'Angers, Angers
  - CH Annecy, Annecy
  - Centre Hospitalier Argenteuil, Argenteuil
  - Centre Hospitalier D'Avignon, Avignon
  - CH Beziers, Béziers
  - Institut Bergonie, Bordeaux
  - Cabinet D'hematologie De La Clinique Du Parc, Castelnau-le-Lez
  - CH William Morey, Chalon-sur-Saône
  - CH Chambery, Chambéry
  - CHU Estaing Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, François Mitterrand, Dijon
  - Centre Hospitalier De Dunkerque, Dunkirk
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - CH De Versailles (Andre Mignot), Le Chesnay
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CH De Libourne, Libourne
  - CHRU De Lille - Hôpital Huriez, Lille
  - CH Limoges, Limoges
  - Leon Berard, Lyon, Lyon
  - Centre Hospitalier De Meaux, Meaux
  - Hopitaux Prives Metz Centre De Belle-Isle, Metz
  - CH De Metz (Hopital De Mercy - CHR Metz Thionville), Metz
  - CHU Montpellier, Montpellier
  - Hopital Salpetriere, Paris
  - La Pitié Salpêtrière - Paris, Paris
  - Hopital Necker, Paris
  - CH St Jean, Perpignan
  - CHU De Poitiers, Poitiers
  - Hôpital Rene Dubos, Pontoise
  - CH De Cornouaille, Quimper
  - CHU De Rennes, Rennes
  - Hopital Victor Provo, Roubaix
  - La Clinique Sainte-Anne, Strasbourg
  - CHRU Strasbourg, Strasbourg
  - Institut Universitaire Du Cancer Toulouse - Oncopo, Toulouse
  - CH Troyes, Troyes
  - CHRU De Nancy - Hôpitaux De Brabois, Vandœuvre-lès-Nancy
  - CHU Sud, St Pierre - La Réunion, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huguet F, Guerci-Bresler A, Roth-Guepin G, Cayssials E, Slama B, Santagostino A, Penot A, Quittet P, Cony-Makhoul P, Saad A, Bastie JN, Hacini M, Coiteux V, Uzunov M, Roy L, Le Clech L, Berger M, Agneray AM, Messas E, Etienne G, Turhan A, Nicolini FE, Rousselot P. Clinical outcomes in patients in any phase of CML treated with ponatinib in France-Data from the TOPASE observational study. Br J Haematol. 2024 Dec;205(6):2295-2304. doi: 10.1111/bjh.19819. Epub 2024 Nov 6. PMID 39506529